CLINICAL TRIAL: NCT00568373
Title: Gastric Electric Stimulation-Enterra Therapy for the Treatment of Chronic Intractable (Drug Refractory) Nausea and Vomiting Secondary to Gastroparesis of Diabetic or Idiopathic Etiology
Brief Title: Gastric Pacemaker Implantation for Gastroparesis
Acronym: HUD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: this is not a clinical trial and does not require registration
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0705-32
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Gastric electrical stimulator
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Intervention Model Description: All patients who have severe symptoms and have been identified by the PI and Sub I to qualify for the treatment will be under one single group

ARMS (1):
- Treatement (Experimental): All subjects that meet the requirement for gastric stimulator placement
  Interventions: Device: Enterra Gastric Pacemaker

INTERVENTIONS:
Device: Enterra Gastric Pacemaker — Gastric Pacemaker

SUMMARY:
Gastric pacemakers and/or temporary gastric stimulators will be implanted in eligible patients.

DETAILED DESCRIPTION:
Due to HUD status, this protocol is for implant only. This is NOT a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Used only if patients have tried and failed conventional treatment ( drug therapy and dietary modification)due to intractable nausea and vomiting secondary to gastroparesis of diabetic or idiopathic etiology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

IPD SHARING:
Plan to Share IPD: No